CLINICAL TRIAL: NCT02045316
Title: The Expression of Aquaporin 3, 8 and 9 in Placenta, Umbilical Cord and Fetal Membranes in Normal Pregnancies and Pregnancies Complicated by Preeclampsia: Perinatal and Neonatal Outcomes.
Brief Title: The Expression of Aquaporin 3, 8 and 9 in Placenta in Normal and Preeclamptic Pregnancies: Perinatal and Neonatal Outcomes.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rakhshanda Aslanova (Other)
Responsible Party: Sponsor-Investigator, Rakhshanda Aslanova, MD, Trakya University
Organization: Trakya University (Other)
Other Study IDs: RA-221281
Record Dates: First submitted 2013-11-18; First posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Aquaporins; Placenta
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Preeclamptic pregnants: pregnants with preeclampsia
- Normal pregnants: pregnants without obstetric complications

SUMMARY:
The etiologic agent responsible for the development of preeclampsia remains unknown. Aquaporins, members of integral membrane proteins, are responsible of water molecules movements through the plasma membrane channels, energy metabolism and associated with changes in cellular volume during apoptosis.

İn such placental pathology as preeclampsia, characterized with superficial implantation and increased apoptosis leading to a relative hypoxia between mother and fetus, the hypothesis of aquaporins important role in energy homeostasis and apoptosis maybe suggested.

DETAILED DESCRIPTION:
The investigators are carrying out a study of 210 pregnant women , from whom 105 will have pregnancy complicated with preeclampsia and 105 with normal pregnancy.

The investigators aim is to investigate the role of the placenta, umbilical cord and amniotic membrane aquaporin expression in etiopathogenesis of preeclampsia. The investigators will compare aquaporin levels in preeclamptic and normal placentas, umbilical cords and amniotic membranes , and investigate relation between aquaporin levels and perinatal ( maternal blood pressure, proteinuria, maternal-fetal doppler ultrasound, amniotic fluid index, fetal intrauterine growth) and neonatal ( Apgar score, biometry, complications) finding.

ELIGIBILITY:
Inclusion Criteria:

* Preeclamptic pregnants
* Normal non-complicated pregnants

Exclusion Criteria:

-Pregnants with another obstetric complications

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 105 pregnant women with preeclampsia and 105 women with normal pregnancy, who applied to Trakya University Faculty of Medicine's.
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
immunohistochemistry | up to 2 week
  Compare aquaporin levels in normal and preeclamptic placentas

SECONDARY OUTCOMES:
Statistical analysis | up to 2 week
  Correlate aquaporin expression with perinatal and neonatal outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Sayin, Professor, Study Chair — Trakya University
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

REFERENCES:
- [Background] Damiano AE. Review: Water channel proteins in the human placenta and fetal membranes. Placenta. 2011 Mar;32 Suppl 2:S207-11. doi: 10.1016/j.placenta.2010.12.012. Epub 2011 Jan 5. PMID 21208655
- [Background] Damiano AE, Zotta E, Ibarra C. Functional and molecular expression of AQP9 channel and UT-A transporter in normal and preeclamptic human placentas. Placenta. 2006 Nov-Dec;27(11-12):1073-81. doi: 10.1016/j.placenta.2005.11.014. Epub 2006 Feb 9. PMID 16480766
- [Background] Leung DN, Smith SC, To KF, Sahota DS, Baker PN. Increased placental apoptosis in pregnancies complicated by preeclampsia. Am J Obstet Gynecol. 2001 May;184(6):1249-50. doi: 10.1067/mob.2001.112906. PMID 11349196
- [Background] Marino GI, Castro-Parodi M, Dietrich V, Damiano AE. High levels of human chorionic gonadotropin (hCG) correlate with increased aquaporin-9 (AQP9) expression in explants from human preeclamptic placenta. Reprod Sci. 2010 May;17(5):444-53. doi: 10.1177/1933719110361385. Epub 2010 Mar 10. PMID 20220109
- [Background] Castro-Parodi M, Levi L, Dietrich V, Zotta E, Damiano AE. CFTR may modulate AQP9 functionality in preeclamptic placentas. Placenta. 2009 Jul;30(7):642-8. doi: 10.1016/j.placenta.2009.04.012. Epub 2009 May 28. PMID 19481256
- [Background] Damiano A, Zotta E, Goldstein J, Reisin I, Ibarra C. Water channel proteins AQP3 and AQP9 are present in syncytiotrophoblast of human term placenta. Placenta. 2001 Sep-Oct;22(8-9):776-81. doi: 10.1053/plac.2001.0717. PMID 11597198